CLINICAL TRIAL: NCT07187141
Title: Phase I Study of the Safety, Tolerability, and Immune Effects of Nasal Protollin in Subjects With Early Symptomatic Alzheimer's Disease
Brief Title: Nasal Protollin in Early Symptomatic Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: I-Mab Biopharma US Limited (Industry)
Responsible Party: Principal Investigator, Tanuja Chitnis, Senior Neurologist, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021P000774
Record Dates: First submitted 2025-09-02; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer Disease (AD)
Keywords: Alzheimer's disease; Protollin; immune response
MeSH Terms: conditions — Alzheimer Disease | interventions — Protollin

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, Phase I, ascending dose study evaluating four dose cohorts.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A (Active Comparator): Protollin 0.1 mg or placebo
  Interventions: Drug: Protollin
- Cohort B (Active Comparator): Protollin 0.5 mg or placebo
  Interventions: Drug: Protollin
- Cohort C (Active Comparator): Protollin 1.0 mg or placebo
  Interventions: Drug: Protollin
- Cohort D (Active Comparator): Protollin 1.5 mg or placebo
  Interventions: Drug: Protollin

INTERVENTIONS:
Drug: Protollin — For the 0.1, 0.5, and 1.0 mg dose groups, Protollin (450 μL per vial) in an aqueous buffer will be administered in two, 0.1 μL sprays, one per nostril. For the 1.5 mg dose group, Protollin (450 muL per vial) in an aqueous buffer will be administered in three, 0.1 μL sprays, two in one nostril and one in the other nostril.

SUMMARY:
In this research study investigators aim to learn more about a new drug called Protollin as a possible new treatment for Alzheimer's Disease (AD). The primary goal is to assess the safety and tolerability.

DETAILED DESCRIPTION:
In this research study investigators want to learn more about a new drug called nasal Protollin as a possible new treatment for Alzheimer's Disease (AD). In AD, there is accumulation in the brain of a toxic substance called amyloid. It is believed that this toxic substance causes brain cells to progressively waste away (degenerate) and die, causing a continuous decline in thinking, behavioral and social skills. Why amyloid accumulates is not completely understood.

The aim of this treatment is to remove toxic amyloid from the brain and prevent further degeneration. Although nasal Protollin has been given as part of vaccination programs, this is the first time Protollin will be given nasally (through the nose) in AD patients. Investigators aim to see if this way of giving the Protollin is safe and whether it stimulates the body's white blood cells to remove toxic amyloid from the brain and ultimately improve cognition. This will be a dose escalating (gradually increasing the dose in different subjects) study, which means we want to find the highest dose of Protollin that is safe to take. Protollin is not approved by the U.S. Food and Drug Administration (FDA). This means that Protollin can only be used in research studies.

This research study will compare Protollin to placebo. The placebo looks exactly like Protollin, but it does not contain any Protollin. During this study participants may get a placebo instead of Protollin. Placebos are used in research studies to see if the results are due to the study drug or due to other reasons.

ELIGIBILITY:
Inclusion Criteria:

1. The Sponsor will rely on NIA-AA Alzheimer's Disease Diagnostic Guidelines1 for Early Symptomatic Alzheimer's Disease and have a MMSE of 29-20.
2. Age between 60-85 years (inclusive).
3. Good general health with no disease expected to interfere with the study.
4. On a stable medication regimen for 8 weeks prior to the study and which is anticipated to remain stable during the study.
5. Subject is not pregnant, lactating, or of childbearing potential (i.e., women must be two years post-menopausal or surgically sterile). ). If a woman is of childbearing potential, her partner is required to use contraception throughout the study (for those identifying as male).
6. Amyloid-positive PET scan (if subject meets all other inclusion criteria).
7. Ability to understand and provide informed consent.

Exclusion Criteria:

1. Any significant neurologic disease including Parkinson's disease, multi-infarct dementia, Huntington's disease, frontotemporal dementia, Lewy body dementia, normal pressure hydrocephalus, brain tumor, brain hemorrhage with persistent neurologic deficits, progressive supra-nuclear palsy, seizure disorder, multiple sclerosis, or history of significant head trauma followed by persistent neurologic defaults or known structural brain abnormalities.
2. Clinically significant or unstable medical condition, including uncontrolled hypertension, uncontrolled diabetes, or significant cardiac, pulmonary, renal, hepatic, endocrine, or other systemic disease.
3. History of autoimmune disease.
4. Current treatment with immunomodulatory or immunosuppressive drugs, or corticosteroid administration by any route of administration (including nasal corticosteroids) within the past month.
5. Major depression or bipolar disorder or a history of schizophrenia.
6. History of alcohol or substance abuse or dependence within the past 2 years.
7. History within the last 5 years of a primary or recurrent malignant disease with the exception of non-melanoma skin cancers, resected cutaneous squamous cell carcinoma in situ, basal cell carcinoma, cervical carcinoma in situ, or in situ prostate cancer with normal prostate-specific antigen post-treatment.
8. Clinically significant abnormalities (defined as greater than mild on the FDA's vaccine toxicity scale) in screening laboratories.
9. Participation in another clinical trial of an investigational drug concurrently or within the past 30 days.
10. Active COVID-19 disease
11. Amyloid-negative PET scan (at screening)
12. COVID-19 vaccine within past 10 days or any other vaccine within past 7 days (at dosing)

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2023-02-21 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of ascending doses of nasal Protollin | Day 1 (enrollment) to 180 days (end of study)
  Safety and tolerability of ascending doses of nasal Protollin following administration of two doses one week apart in subjects, 60-85 years inclusive with Early Symptomatic Alzheimer's Disease (29-20 MMSE classification). Safety will be assessed by physical examination (including evaluation of the nose and oropharynx), laboratory studies, EKG, and elicited and spontaneously reported signs and symptoms, using the FDA Guidance for Industry: Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (September 2007) for the evaluation of toxicities and reactogenicity. Tolerability will be assessed by the degree of severity of both spontaneously reported and elicited symptoms and associated signs, systemically and at the site of administration following administration of nasal Protollin, if thought by the investigator to be related or possibly related to its administration.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No